CLINICAL TRIAL: NCT06658249
Title: Comparative Effects of Core Stabilization Exercises Versus Foot-Ankle Strengthening Program on Pain, Physical Function and Quality of Life in Patients With Knee Osteoarthritis.
Brief Title: Effects of Core Stabilization Exercises Versus Foot-Ankle Strengthening Program in Patients With Knee Osteoarthritis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0132
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis (OA)
Keywords: Knee Osteoarthritis; Pain; Physical Function; Quality of Life
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Stabilization Exercises with Foot-Ankle Strengthening Program (Experimental): Core Stabilization Exercises with Foot-Ankle Strengthening Program along with simple conventional treatment.
  Interventions: Other: Core Stabilization Exercises with Foot-Ankle Strengthening Program
- Foot-Ankle Strengthening Program (Active Comparator): Foot-Ankle Strengthening Program along with simple conventional treatment
  Interventions: Other: Foot-Ankle Strengthening Program

INTERVENTIONS:
Other: Core Stabilization Exercises with Foot-Ankle Strengthening Program — Core Stabilization Exercises and Foot-Ankle Strengthening Program with the frequency of 3 sets of 10 repetitions 3 times per week for a total duration of 6 weeks. Core Stabilization Exercises include : Double leg Abdominal Press, Single Leg Abdominal Press, Abdominal crunches, Side-lying Hip Abduction, Bridging Exercise, Wall Squats Exercise. Foot-Ankle Strengthening Program include : Step ups Exercise, Heel Raises in standing/sitting, Toe Raises in standing/sitting, Foot-Ankle isometrics with theraband, One leg balance with chair support. Pre and Post intervention values will be taken on 1st day and after 6 weeks. Simple Conventional treatment will also given that include Hot Pack and TENS for 10 minutes and Ultrasound for 5 minutes and Knee Isometric exercises with the frequency of 1 set of 10 repetitions with 5 sec hold with the ratio of 3 times per week for a total duration of 6 weeks.
  Other Names: Simple Conventional Treatment
  Arms: Core Stabilization Exercises with Foot-Ankle Strengthening Program
Other: Foot-Ankle Strengthening Program — Foot-Ankle Strengthening Program along with common conventional treatment with the frequency of 3 sets of 10 repetition thrice per week for a total duration of 6 weeks. Core Stabilization Exercises include : Double leg Abdominal Press, Single Leg Abdominal Press, Abdominal crunches, Side-lying Hip Abduction, Bridging Exercise, Wall Squats Exercise. Foot-Ankle Strengthening Program include : Step ups Exercise, Heel Raises in standing/sitting, Toe Raises in standing/sitting, Foot-Ankle isometrics with theraband, One leg balance with chair support. Pre and Post intervention values will be taken on 1st day and after 6 weeks. Simple Conventional treatment will also given that include Hot Pack and TENS for 10 minutes and Ultrasound for 5 minutes and Knee Isometric exercises with the frequency of 1 set of 10 repetitions with 5 sec hold with the ratio of 3 times per week for a total duration of 6 weeks.
  Other Names: Simple Conventional Treatment
  Arms: Foot-Ankle Strengthening Program

SUMMARY:
Knee osteoarthritis (OA) is also known as degenerative joint disease, is typically the result of wear and tear and progressive loss of articular cartilage. It is most common in the elder population. It results from functional disability and altered knee biomechanics. Risk factors of Knee OA include; older age, genetics and obesity, female gender. The aim of this study is to compare the effects of core stabilization exercises versus foot-ankle strengthening program on pain, physical function and quality of life in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
A Randomized Clinical Trial will be conducted at Riphah Physiotherapy Clinic Lahore, FMH Physiotherapy Department, Hamza Hospital Physiotherapy Clinic, Lahore through convenient purposive sampling technique 46 patients which will be allocated by using simple randomization through computer generated software into Group A and Group B. Group A will be treated with core stabilization exercises and ankle-foot strengthening program and Group B will be treated with ankle-foot strengthening program at the frequency of 3 sets with 10 repetitions thrice per week in the total duration of 6 weeks. Outcome measures will be conducted through (NPRS), (WOMAC), Knee Osteoarthritis Outcome Score (KOOS) Questionnaire and quality of life (SF-36) questionnaire before and after 6 weeks. Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Both genders of 40-65 years of age will include in this study.
* Knee OA of grade 1-2.
* Individuals with significant unilateral and bilateral knee osteoarthritis. symptoms and positive radio-graphical findings.
* Difficulty in walking/stair climbing.

Exclusion Criteria:

* Any history of knee fracture/ tumor/ infection and hip/knee surgery.
* Total Knee Replacement patients.
* Neurological disease.
* Patient received physical therapy treatment from last 6 months.
* Inflammatory Arthritis (Rheumatoid Arthritis)
* Use of any intra-articular injections (steroid/ hyaluronic acid/ PRP.) from last 3-6 months.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-01-07 (Estimated); Study Completion 2025-01-07 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 6 weeks
  Changes from baseline, Numeric Rating Scale (NRS) is the most commonly used scale in which the pain rate ranges from 0 (no pain) to 10 (worst pain). The level of knee perception of pain is assessed by using the NPRS. It is used as the outcome measure tool for patients with OA knee. The NPRS is consider as reliable, valid, and responsive scale for pain. This scale has high reliability (0.95-0.96).
  The validity of NPRS ranges from (0.86-0.95).
Knee Injury and Osteoarthritis Outcome Score (KOOS) Questionnaire | 6 weeks
  Changes from baseline, KOOS score consist of five patient-relevant dimensions that are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. This scale consist of total 42-items and score of this scale range from 0 (severe knee pathology) to 100 (no knee problem). This tool has been use to assess the pain, symptoms, activities level, function in knee osteoarthritis patients. It is a valid tool for Knee Osteoarthritis patients ; validity ranges up-to (0.80-0.89).
WESTREN ONTARIO AND MCMASTER UNIVERSITIES OSTEOARTHRITIS INDEX (WOMAC SCALE) | 6 weeks
  Changes from baseline, WOMAC scale consist of three subscales: pain (five questions), stiffness (two questions), and physical function (17 questions). The subscale scores can vary, with pain ranging from 0 to 20 points; stiffness, 0 to 8 points; and physical function, 0 to 68 points. Higher scores have been represent worse pain, stiffness, and functional limitations. This scale will be use to assess pain, stiffness, physical function level in knee osteoarthritis patients.
36- Items Short Form Survey (SF-36) QUESTIONNAIRE | 6 weeks
  Changes from baseline, Quality of life scale (SF-36) questionnaire consist of subscale of general health, activities limitations, physical health problems, emotional health problems, social activities, energy and emotions; total 36 items in it. SF-36 is used to assess the quality of life in knee osteoarthritis patient. SF-36 questionnaire is reliable and valid tool for quality of life in knee osteoarthritis individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Fatima Memorial Hospital Physical Therapy Department, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oiestad BE, Aroen A, Rotterud JH, Osteras N, Jarstad E, Grotle M, Risberg MA. The efficacy of strength or aerobic exercise on quality of life and knee function in patients with knee osteoarthritis. A multi-arm randomized controlled trial with 1-year follow-up. BMC Musculoskelet Disord. 2023 Sep 8;24(1):714. doi: 10.1186/s12891-023-06831-x. PMID 37684597
- [Background] Holm PM, Schroder HM, Wernbom M, Skou ST. Low-dose strength training in addition to neuromuscular exercise and education in patients with knee osteoarthritis in secondary care - a randomized controlled trial. Osteoarthritis Cartilage. 2020 Jun;28(6):744-754. doi: 10.1016/j.joca.2020.02.839. Epub 2020 Mar 13. PMID 32179197
- [Background] Hernandez D, Dimaro M, Navarro E, Dorado J, Accoce M, Salzberg S, Policastro PO. Efficacy of core exercises in patients with osteoarthritis of the knee: A randomized controlled clinical trial. J Bodyw Mov Ther. 2019 Oct;23(4):881-887. doi: 10.1016/j.jbmt.2019.06.002. Epub 2019 Jun 4. PMID 31733777
- [Background] GBD 2021 Osteoarthritis Collaborators. Global, regional, and national burden of osteoarthritis, 1990-2020 and projections to 2050: a systematic analysis for the Global Burden of Disease Study 2021. Lancet Rheumatol. 2023 Aug 21;5(9):e508-e522. doi: 10.1016/S2665-9913(23)00163-7. eCollection 2023 Sep. PMID 37675071